CLINICAL TRIAL: NCT03560050
Title: Compliance and Technical Assistance for Child and Adult Care Food Program in Family Child Care Homes
Brief Title: Technical Assistance for Child and Adult Care Food Program in Family Child Care Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Susan B. Sisson, Associate Professor, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7551
Record Dates: First submitted 2018-05-23; First posted 2018-06-18 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Nutrition Poor; Health Behavior
Keywords: early childhood education; family child care home; food environment
MeSH Terms: conditions — Malnutrition; Health Behavior | interventions — Food Assistance

STUDY DESIGN:
Intervention Model Description: Randomized trial where family child care home providers (the participant) are randomized to either nutrition or environmental health technical assistance intervention. Interventions are matched for time and contact
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Nutrition assistance (Experimental): three encounters with Intervention team over three months: two home-based visits for 90 minutes each scheduled at the convenience of the provider and a 3- hour group class session with other providers.
  Interventions: Behavioral: Nutrition assistance
- Behavioral: Children's environmental health (Experimental): three encounters with Intervention team over three months: two home-based visits for 90 minutes each scheduled at the convenience of the provider and a 3- hour group class session with other providers.
  Interventions: Behavioral: Children's environmental health

INTERVENTIONS:
Behavioral: Nutrition assistance — Participating family child care home providers in and around the Oklahoma City (OKC) area will be randomized to either the Nutrition (n=26), or an environmental health comparison group (n=26). Briefly, the Nutrition Technical Assistance Intervention and comparison group will consist of three encounters with the intervention team: two home-based, 90-minute visits scheduled at the convenience of the family child care home provider and a 3-hour group class session that will be conducted on a weekend. Total contact time with intervention staff will be 6 hours. All participants will receive a toolkit. Providers will complete either intervention over a period of three months.
  Arms: Behavioral: Nutrition assistance
Behavioral: Children's environmental health — Participating family child care home providers in and around the OKC area will be randomized to either the Nutrition (n=26), or an environmental health intervention (n=26) that will receive an Integrated Pest Management and Green Cleaning intervention with the same format and visit frequency. Briefly, the Intervention will consist of three encounters with the intervention team: two home-based, 90-minute visits scheduled at the convenience of the family child care home provider and a 3-hour group class session that will be conducted on a weekend. Total contact time with intervention staff will be 6 hours. All participants will receive a toolkit. Providers will complete either intervention over a period of three months.
  Arms: Behavioral: Children's environmental health

SUMMARY:
This study evaluates the effect of a nutrition technical assistance training program for family child care home providers on the food they serve young children in their care and the food environment in their home. Half the providers will be assigned to the nutrition program and the other half will receive a comparison on environmental health.

DETAILED DESCRIPTION:
Early care and education (ECE) providers play a vital role in ensuring that young children have access to nutritious foods. Over 25% of children in ECE (1.2 million children) attend Family Child Care Homes (FCCH). Improvements in the Child and Adult Care Food Program (CACFP) may introduce new barriers for FCCH, which have limited meal preparation capacity. Limited research has examined foods served by FCCH providers, and no group randomized trials have been conducted using a Community-Based Participatory approach in FCCH and including an evaluation of intervention costs.

Goals: 1. Determine compliance of menus and meals provided in FCCH with CACFP guidelines. 2. Determine the effectiveness of a pilot community-based Nutrition Technical Assistance intervention to enhance meeting CACFP best-practices. 3. Determine the effectiveness of a statewide community-based Nutrition Technical Assistance Intervention to enhance meeting CACFP best-practices. 4. Expand university student opportunities for participation in health research.

Methods: Conduct a cross-sectional assessment of a random sample of FCCH providers' (n=52) menus and meals served. Foods will be evaluated against the CACFP requirements and best-practices. After the cross-sectional examination, providers in the pilot will be randomly assigned to a Nutrition Technical Assistance (n=26) or attention comparison intervention (n=26). Following the pilot, trained Extension Educators will implement both interventions (n=27 intervention, n=27 comparison) in six selected counties, reaching underserved rural and low-income populations. The intervention is based on theoretical foundations and formative interviews, and will consist of two 60-90-minute visits to the FCCH and one group class lasting approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Family child care home providers within 60 minutes of Oklahoma City who participate in the Child and Adults Care Food Program

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in self-reported nutrition practices | baseline, post 3-months, post 12-months
  Providers report the frequency of fruit and vegetables, milk, and salty snacks served

SECONDARY OUTCOMES:
Change in Provider knowledge and self efficacy | baseline, post 3-months, post 12-months
  providers will self report nutrition and environmental health knowledge and self efficacy
Change in Environmental health observation | baseline, post 3-months, post 12-months
  observation of household cleaners and chemicals and signs of pests
Change in nutrition environment using the Environment and Policy Assessment Observation | baseline, post 3-months, post 12-months
  observation of food environment during lunch on 2 unannounced days
Change in compliance of menu and meal with Child and Adult Care Food Program | baseline, post 3-months, post 12-months
  menus and meals are compared to the requirements and best practices of the CACFP
Change in children's dietary intake | baseline, post 3-months, post 12-months
  observation of children's dietary intake on 2 unannounced days

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Sisson, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Sisson SB, Leidner J, Hall S, Williams BD, Vesely SK, Poe T, Ward DS, Crosscut C, Hildebrand D, Salvatore AL. Three- and Twelve-Month Changes in Child and Adult Care Food Program Best Practices and Preschool Children's Dietary Intake in Family Child Care Homes after the Happy Healthy Homes Randomized Controlled Trial. Child Obes. 2025 Jul;21(5):476-488. doi: 10.1089/chi.2024.0361. Epub 2025 Mar 10. PMID 40059639
- [Derived] Sisson SB, Eckart E, Williams BD, Patel SM, Kracht CL, Davis HA, Ward DS, Hildebrand D, Stoner JA, Stinner E, Kerr KE, Salvatore A. Family child care home providers' self-reported nutrition and physical activity practices, self-efficacy, barriers and knowledge: baseline findings from happy healthy homes. Public Health Nutr. 2022 Aug;25(8):2111-2124. doi: 10.1017/S1368980022000337. Epub 2022 Feb 7. PMID 35125128
- [Derived] Sisson SB, Salvatore AL, Hildebrand D, Poe T, Merchant C, Slawinski M, Kracht CL, Stoner JA, Alcala Lazarte N, Schneider LAF, Weber J, Jones F, Ward D. Interventions to promote healthy environments in family child care homes in Oklahoma-Happy Healthy Homes: study protocol for a randomized controlled trial. Trials. 2019 Aug 30;20(1):541. doi: 10.1186/s13063-019-3616-9. PMID 31470886